CLINICAL TRIAL: NCT00205751
Title: International, Multi-center, Prospective, Double Randomized, Open Phase III Study Evaluating Thalidomide/Dexamethasone Versus Melphalan/Prednisone as Induction Therapy and Thalidomide/Interferon-alpha Versus Interferon-alpha as Maintenance Therapy in Newly Diagnosed Patients With Multiple Myeloma
Brief Title: Thalidomide/Dexamethasone vs MP for Induction Therapy and Thalidomide/Intron A vs Intron A for Maintenance Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Austrian Forum Against Cancer (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-002-0601
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; first line treatment; thalidomide; melphalan
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide/Dexamethasone vs Melphalan/Prednisone

SUMMARY:
This is an international multi-center prospective, double randomized, open, controlled phase III study with a phase II entrance phase to compare the therapeutic efficacy of thalidomide plus dexamethasone to conventional melphalan plus prednisone in newly diagnosed myeloma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Multiple Myeloma of IgG, IgA, IgD, IgE, IgM lambda or kappa light chain, low secretory or non-secretory disease
* WHO performance status 0,1,2,or 3
* No prior treatment of multiple myeloma
* Clear requirement of treatment (usually Durie/Salmon stage II or III)
* Anticipated life expectancy of at least 3 months
* Adequate organ function
* Minimum recovery period of 2 weeks following any major surgical procedure before entry into this study
* Women, who are sterilized via hysterectomy or bilateral tubal ligation or at least one year post-menopausal
* Age of at least 19 years, there is no upper age limit patients must have been informed and must have signed an informed consent

Exclusion Criteria:

* Extramedullary plasmocytoma or solitary plasmocytoma without evidence of dissemination of disease
* Benign monoclonal gammopathy
* Multiple myeloma of IgM without osteolytic bone lesions
* Smouldering myeloma
* More than 3 irradiation fields
* Irreversible performance status of WHO4
* Prior treatment of myeloma with any of the following: chemotherapeutic or immunomodulatory agents, corticosteroids, antiangiogenic agents or other investigational drugs
* Women of childbearing potential
* Preexisting peripheral polyneuropathy
* Congestive heart failure NYHA III, IV
* Acute infection requiring systemic antibiotics at study entry until resolved
* Any uncontrolled underlying medical condition (eg diabetes, glaucoma)
* Second primary malignancy (with the exception of cervical carcinoma in situ and non-myeloma skin malignancies) unless patient has been disease-free for at least three years

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2001-08; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Time to progression
Response rate

SECONDARY OUTCOMES:
Survival
Time to response
Toxicity
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Ludwig, MD,Univ.Prof, Principal Investigator — Wilhelminenspital 1st medical dep.-center for oncology and hematology
Locations (1):
- Wilhelminenspital, 1st Medical Department-center for oncology and hematology, Vienna, Austria

REFERENCES:
- [Derived] Ludwig H, Adam Z, Tothova E, Hajek R, Labar B, Egyed M, Spicka I, Gisslinger H, Drach J, Kuhn I, Hinke A, Zojer N. Thalidomide maintenance treatment increases progression-free but not overall survival in elderly patients with myeloma. Haematologica. 2010 Sep;95(9):1548-54. doi: 10.3324/haematol.2009.020586. Epub 2010 Apr 23. PMID 20418244
- [Derived] Ludwig H, Hajek R, Tothova E, Drach J, Adam Z, Labar B, Egyed M, Spicka I, Gisslinger H, Greil R, Kuhn I, Zojer N, Hinke A. Thalidomide-dexamethasone compared with melphalan-prednisolone in elderly patients with multiple myeloma. Blood. 2009 Apr 9;113(15):3435-42. doi: 10.1182/blood-2008-07-169565. Epub 2008 Oct 27. PMID 18955563